CLINICAL TRIAL: NCT03218917
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Center Study to Assess the Efficacy, Safety & Tolerability, and PK of INS1007 Administered Once Daily for 24 Weeks in Subjects With Non-CF Bronchiectasis - The Willow Study
Brief Title: Assessment of INS1007 in Participants With Non-Cystic Fibrosis Bronchiectasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INS1007-201; 2017-002533-32 (EudraCT Number)
Record Dates: First submitted 2017-07-11; First posted 2017-07-17 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Non-Cystic Fibrosis Bronchiectasis
Keywords: P aeruginosa; bronchiectasis; active neutrophil elastase
MeSH Terms: conditions — Bronchiectasis | interventions — brensocatib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Brensocatib 10 mg (Experimental): Participants received brensocatib 10 mg once daily (QD) before breakfast, for 24 weeks.
  Interventions: Drug: Brensocatib 10 mg
- Brensocatib 25 mg (Experimental): Participants received brensocatib 25 mg QD before breakfast, for 24 weeks.
  Interventions: Drug: Brensocatib 25 mg
- Placebo (Placebo Comparator): Participants received the matching placebo QD before breakfast, for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brensocatib 10 mg — Administered once per day for 24 weeks
  Arms: Brensocatib 10 mg
Drug: Brensocatib 25 mg — Administered once per day for 24 weeks
  Arms: Brensocatib 25 mg
Drug: Placebo — Administered once per day for 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate if INS1007 can reduce pulmonary exacerbations over a 24-week treatment period in participants with non-cystic fibrosis bronchiectasis.

DETAILED DESCRIPTION:
Phase 2 randomized, double-blind, placebo-controlled, parallel-group, multicenter, multi-national study to assess the efficacy, safety and tolerability, and pharmacokinetics (PK) of INS1007 administered once daily for 24 weeks in participants with non-cystic fibrosis bronchiectasis (NCFBE).

ELIGIBILITY:
Inclusion Criteria:

1. Clinical history consistent with NCFBE (cough, chronic sputum production and/or recurrent respiratory infections)
2. Are current sputum producers with a history of chronic expectoration and able to provide a sputum sample during Screening
3. Have at least 2 documented pulmonary exacerbations in the past 12 months before Screening

Exclusion Criteria:

1. Have a primary diagnosis of chronic obstructive pulmonary disease (COPD) or asthma
2. Have bronchiectasis due to cystic fibrosis (CF), hypogammaglobulinemia, common variable immunodeficiency, or alpha1-antitrypsin deficiency
3. Are current smokers
4. Are currently being treated for a nontuberculous mycobacterial lung infection, allergic bronchopulmonary aspergillosis, or tuberculosis
5. Have any acute infections, (including respiratory infections)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Fernandez, MD, Study Director — Insmed Incorporated
Locations (108):
- United States (36):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Medical Group, Peoria, Arizona
  - NewportNativeMD, Newport Beach, California
  - Palmtree Clinical Research, Palm Springs, California
  - UC Davis Medical Center, Sacramento, California
  - Stanford University Medical Center, Stanford, California
  - National Jewish Heath, Denver, Colorado
  - UConn Health Center, Farmington, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Clinical Research Specialists, LLC, Celebration, Florida
  - St. Francis Medical Institute, Clearwater, Florida
  - University of Florida, Gainesville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Sarasota Memorial Hospital Clinical Research Center, Sarasota, Florida
  - The Emory Clinic, Pulmonology, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - LSU Health Sciences Center, New Orleans, Louisiana
  - Johns Hopkins University, Division of Pulmonary and Critical Care Medicine, Baltimore, Maryland
  - Pulmonary and Critical Care Associates of Baltimore, Towson, Maryland
  - Mid Atlantic Pulmonary & Research Center, Westminster, Maryland
  - Michigan Medicine, Ann Arbor, Michigan
  - NYU Pulmonary & Critical Care Associates, New York, New York
  - Columbia University Medical Center/ New York Presbyterian Hospital, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Novant Health Pulmonary Medicine South, Charlotte, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - SMS Clinical Research, LLC, Mesquite, Texas
  - The University of Texas Health Science at Tyler, Tyler, Texas
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
- Australia (9):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Mater Misericordia Medical Centre, Brisbane, Queensland
  - Gallipoli Medical Research Foundation, Brisbane, Queensland
  - Metro North Hospital and Health Service (The Prince Charles Hospital), Chermside, Queensland
  - Respiratory Clinical Trials Unit, Royal Adelaide Hospital, Adelaide, South Australia
  - Respiratory Clinical Trials PTY LTD, Kent Town, South Australia
  - Box Hill Hospital, Eastern Clinical Research Unit, Box Hill, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Institute for Respiratory Health, Nedlands, Western Australia
- UZ Leuven, Leuven, Vlaams Brabant, Belgium
- Bulgaria (4):
  - Medical Center ReSpiro Ltd (Kiselov), Razgrad, Momina
  - Medical Center UNIMED, Plovdiv
  - MHAT "Dr IvanSeliminski"-Sliven, Sliven
  - Cardioart Medical Center, Stara Zagora
- Denmark (3):
  - Hvidovre Hospital, Hvidovre, Capital Region
  - Aarhus University Hospital, Aarhus
  - Sjællands Universitetshospital, Roskilde, Roskilde
- Germany (10):
  - Krankenhaus Donaustauf, Donaustauf, Bavaria
  - Klinikum der Universität München Medizinische Klinik V Pneumologie / Mukoviszidose-Zentrum für Erwachsene, Munich, Bavaria
  - Klinikum Nuernberg, Nuremberg, Bavaria
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - IKF Pneumologie Frankfurt, Frankfurt am Main, Hesse
  - Ruhrlandklinik Essen, University Essen, Essen, North Rhine-Westphalia
  - Forschungszentrum Borstel, Borstel, Schleswig-Holstein
  - Universitätsklinikum Jena, Jena, Thuringia
  - Research Center for Medical Studies (RCMS), Berlin
  - Städt. Klinikum München GmbH, Bogenhausen, München
- Italy (5):
  - University of Milan, IRCCS Fondazione Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Ospedale San Gerardo, Monza, Monza E Brianza
  - University Hospital of Pisa, Pisa, Via Paradisa 2
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - ICS Maugeri spa SB, IRCSS Telese, Telese Terme
- Netherlands (4):
  - Noordwest Ziekenhuis Group, Alkmaar
  - Amphia Longresearch Astma/COPD Uni 52/5e etage, Breda
  - RadboudUMC, location Dekkerswald, Nijmegen
  - Zuyderland MC, Sittard
- New Zealand (5):
  - P3 Research, Tauranga, BOP
  - P3 Research (Hawke's Bay), Hastings, Hawkes Bay
  - Southern District health Board/Dunedin Hospital, Dunedin, Otago
  - Waikato District Health Board, Hamilton, Waikato Region
  - Auckland District Health Board, Greenlane clinical Centre, Auckland
- Poland (5):
  - Centrum Badan Klinicznych, Piotr Napora Lekarze i Spolka Partnerska, Osrodek Badan Wczesnej Fazy, Wroclaw, Lower Silesian Voivodeship
  - Grażyna Jasieniak Pinis Niepubliczny Zakład Opieki Zdrowotnej Atopia, Krakow
  - NZOZ Krak-Medyk Sp. z o.o, Krakow
  - Medical University of Lodz Poland, Lodz
  - Gabinet Lekarski Pediatryczno-Alergologiczny Zenon Bukowczan, Sucha Beskidzka
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Changi General Hospital, Singapore
- South Korea (9):
  - Inha University Hospital, Incheon, Jung-gu
  - Gachon University Gil Medical Center, Incheon, Namdong-gu
  - Chonnam National University Hospital, Gwangju
  - The Catholic University of Korea Incheon St. Mary's Hospital, Incheon
  - The Catholic University of Korea, St. Paul's Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (5):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona
  - Hospital Universiatrio y politecnico La Fe, Valencia
- United Kingdom (10):
  - NHS Tayside, Dundee, Angus
  - Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool, Lancashire
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool, Merseyside
  - NHS Lothian, Edinburgh, Scotland
  - Ashford and St Peter's Hospitals NHS Foundation Trust, Chertsey, Surrey
  - The Royal Wolverhampton NHS Trust, Wolverhampton, West Midlands
  - Royal Brompton & Harefield NHS Foundation Trust, London
  - Pennine Acute Hospitals NHS Trust, Manchester
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnson ED, Long MB, Perea L, Shih VH, Fernandez C, Teper A, Cipolla D, McIntosh E, Galloway R, Eke Z, Shuttleworth M, Hull R, Spinou A, De Soyza A, Ringshausen FC, Goeminne P, Lorent N, Haworth C, Loebinger MR, Blasi F, Shteinberg M, Aliberti S, Polverino E, Sibila O, Shoemark A, Mange K, Huang JTJ, Stobo J, Chalmers JD. Broad Immunomodulatory Effects of the Dipeptidyl Peptidase-1 Inhibitor Brensocatib in Bronchiectasis: Data from the Phase 2, Double-Blind, Placebo-controlled WILLOW Trial. Am J Respir Crit Care Med. 2025 May;211(5):770-778. doi: 10.1164/rccm.202408-1545OC. PMID 39938076
- [Derived] Basso J, Chen KJ, Zhou Y, Mark L, LaSala D, Dorfman A, Atalla M, Chun D, Viramontes V, Chang C, Leifer F, McDonald PP, Cipolla DC. The pharmacokinetic profile of brensocatib and its effect on pharmacodynamic biomarkers including NE, PR3, and CatG in various rodent species. Front Pharmacol. 2023 Jul 19;14:1208780. doi: 10.3389/fphar.2023.1208780. eCollection 2023. PMID 37538173
- [Derived] Cipolla D, Zhang J, Korkmaz B, Chalmers JD, Basso J, Lasala D, Fernandez C, Teper A, Mange KC, Perkins WR, Sullivan EJ. Dipeptidyl peptidase-1 inhibition with brensocatib reduces the activity of all major neutrophil serine proteases in patients with bronchiectasis: results from the WILLOW trial. Respir Res. 2023 May 17;24(1):133. doi: 10.1186/s12931-023-02444-z. PMID 37198686
- [Derived] Chalmers JD, Haworth CS, Metersky ML, Loebinger MR, Blasi F, Sibila O, O'Donnell AE, Sullivan EJ, Mange KC, Fernandez C, Zou J, Daley CL; WILLOW Investigators. Phase 2 Trial of the DPP-1 Inhibitor Brensocatib in Bronchiectasis. N Engl J Med. 2020 Nov 26;383(22):2127-2137. doi: 10.1056/NEJMoa2021713. Epub 2020 Sep 7. PMID 32897034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the trial at 116 sites in 14 countries from 31 October 2017 to 12 December 2019.
Pre-assignment Details: 416 participants were screened with 160 participants resulting in a screen failure. A total of 256 participants were randomized.
Groups:
- Brensocatib 10 mg: Participants received brensocatib 10 mg QD before breakfast, for 24 weeks.
Period: Overall Study
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg | Placebo
Started (Intent-to-treat (ITT) population included all the participants who were randomized.) | 82 | 87 | 87
Received Study Treatment (Safety Population) (Safety population included all participants who received at least 1 dose of the study drug.) | 81 | 89 (2 participants, each randomized to placebo and Brensocatib 10 mg, received Brensocatib 25 mg. Both participants were included as randomized in the ITT population and in the INS1007 25 mg group in the Safety population.) | 85
Participants Did Not Receive Drug | 0 | 0 | 1
Pharmacodynamic (PD) Population (PD population included participants who received at least 1 dose of the study drugs, have at least 1 pre-dose and 1 post-dose measurement for neutrophil elastase (NE), or proteinase 3, or cathepsin G, or other biomarkers, and have no major protocol deviations that considered to impact on the analysis of the PD data.) | 80 | 89 | 84
Completed | 76 | 75 | 74
Not Completed | 6 | 12 | 13
Not completed — Adverse Event | 3 | 3 | 2
Not completed — Subject withdrew consent | 2 | 4 | 10
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Reason Missing | 0 | 2 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Non-Compliance with Study Drug | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT population included all the participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg | Placebo | Total
Number analyzed (Participants) | 82 | 87 | 87 | 256
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (12.42) | 63.7 (12.67) | 64.0 (11.86) | 64.1 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 62 | 55 | 174
  Male | 25 | 25 | 32 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 0 | 6
  Not Hispanic or Latino | 80 | 83 | 87 | 250
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian (White) | 76 | 78 | 71 | 225
  Race: African American/Black of African origin | 0 | 2 | 2 | 4
  Race: Asian | 5 | 5 | 13 | 23
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 3
  Race: Other | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to the First Pulmonary Exacerbation Over 24-Week Treatment Period
Description: Time to first pulmonary exacerbation was calculated as the number of days from the date of randomization to the date of first documentation of an exacerbation. Pulmonary exacerbation was defined as having 3 or more of the following symptoms for at least 48 hours resulting in a physician's decision to prescribe antibiotics: 1. Increased cough 2. Increased sputum volume or change in sputum consistency 3. Increased sputum purulence 4. Increased breathlessness and/or decreased exercise tolerance 5. Fatigue and/or malaise 6. Hemoptysis A minimum of 4 weeks must have occurred between one exacerbation onset and the next. Any exacerbation that occurred less than 4 weeks from the prior exacerbation was not considered a new exacerbation. The analysis was performed using the stratified log rank test and using Kaplan Meier (KM) curves.
Time Frame: Baseline (Day 1) to Week 24
Population: ITT population included all participants who were randomized. Overall number of participants analyzed are number of participants with at least one exacerbation over 24-week treatment period.
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg | Placebo
Number analyzed (Participants) | 26 | 29 | 42
days | NA [NA to NA] — The median, upper and lower limit of confidence interval (CI) was not estimated due to insufficient number of participants with exacerbations in Brensocatib 10 mg group. | NA [NA to NA] — The median, upper and lower limit of CI was not estimated due to insufficient number of participants with exacerbations in Brensocatib 25 mg group. | 189.0 [141.0 to NA] — The upper limit of CI was not estimated due to insufficient number of participants with exacerbations in placebo.
Statistical Analysis 1: Comparison: Brensocatib 10 mg; Test type: Superiority; p = 0.014, Stratified Log-rank test — P-value is one-sided for superiority; Stratified by Pseudomonas aeruginosa (Pa) colonization status and maintenance antibiotic use at Baseline
Statistical Analysis 2: Comparison: Brensocatib 25 mg vs Placebo; Test type: Superiority; p = 0.022, Stratified Log-rank test — P-value is one-sided for superiority; Stratified by colonization status and maintenance antibiotic use at Baseline

2. Secondary Outcome: Change From Baseline in Quality of Life Questionnaire - Bronchiectasis (QOL-B) Respiratory Symptoms Domain Score Over 24 Week Treatment Period
Description: The QOL-B is a validated, self-administered patient reported outcome (PRO) that assesses symptoms, functioning, and health-related (HR) QOL for participants with non-cystic fibrosis bronchiectasis (NCFBE). The QOL-B contains 37 items in 8 domains (Respiratory Symptoms, Physical Functioning, Role Functioning, Emotional Functioning, Social Functioning, Vitality, Health Perceptions and Treatment Burden). Each of the 37 items is scored from 1 to 4, and each of the 8 domains scale scores is standardized on a 0-100 point scale, with higher scores representing fewer symptoms or better functioning and HR QoL. A positive change from Baseline indicates improvement in symptoms. For this outcome measure, change in the respiratory symptoms domain score from Baseline was reported. The analysis was based on mixed model for repeated measures (MMRM) approach.
Time Frame: Baseline (Day 1) to Week 24
Population: ITT population included all participants who were randomized. Overall number of participants analyzed are the number of participants with data available for analyses at the latest assessment visit over the 24-week treatment period.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg | Placebo
Number analyzed (Participants) | 75 | 77 | 72
score on a scale | 3.8 (0.78) | 5.9 (0.76) | 5.7 (0.77)

3. Secondary Outcome: Change From Screening in Post-Bronchodilator Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) Over 24-Week Treatment Period
Description: FEV1 was used to assess lung function and is the maximum amount of air that can be forced out in one second after taking a deep breath. The percent predicted FEV1 was calculated by converting the spirometer reading to a percentage of what would be predicted as normal FEV1 based on a several personal factors (e.g. sex, age, etc.). Change from screening in percent predicted FEV1 to Week 24 was calculated as: percent predicted FEV1 value at Week 24 and percent predicted FEV1 value at screening. A positive percent change from screening indicates an improvement in lung function. The analysis was done using analysis of covariance (ANCOVA) with Pa colonization status and maintenance macrolide antibiotic use at Baseline as covariates.
Time Frame: Screening (Days -42 to -1) to Week 24
Population: ITT population included all participants who were randomized. Overall number of participants analyzed are the number of participants with data available for analyses over the 24-week treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent predicted FEV1
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg | Placebo
Number analyzed (Participants) | 77 | 77 | 73
percent predicted FEV1 | -0.3 (0.88) | -0.3 (0.85) | -1.8 (0.87)

4. Secondary Outcome: Change From Baseline in Concentration of Active Neutrophil Elastase (NE) in Sputum
Description: The concentration of active NE in sputum, was measured by the difference between the pre-treatment concentration and on-treatment concentration. In bronchiectasis, activation of neutrophils in the airway leads to release of NE which leads to damaged airway walls, mucus hypersecretion, exacerbated inflammation, which in turn affects neutrophil and macrophage functions, increasing the risk of infection. Negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 24
Population: Pharmacodynamic population included participants who received at least 1 dose of the study drugs, have at least 1 pre-dose and 1 post-dose measurement for NE, or proteinase 3, or cathepsin G, or other biomarkers, and have no major protocol deviations that considered to impact on the analysis of the PD data.
Measure: Least Squares Mean (Standard Error); unit: microgram/ milliliter (µg/mL)
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg | Placebo
Number analyzed (Participants) | 80 | 89 | 84
microgram/ milliliter (µg/mL) | -2.928 (0.351) | -4.117 (0.322) | -1.409 (0.313)

5. Secondary Outcome: Number of Participants Who Experienced a Pulmonary Exacerbation
Description: Pulmonary exacerbation was defined as having 3 or more of the following symptoms for at least 48 hours resulting in a physician's decision to prescribe antibiotics. 1. Increased cough 2. Increased sputum volume or change in sputum consistency 3. Increased sputum purulence 4. Increased breathlessness and/or decreased exercise tolerance 5. Fatigue and/or malaise 6. Hemoptysis A minimum of 4 weeks must have occurred between one exacerbation onset and the next. Any exacerbation that occurred less than 4 weeks from the prior exacerbation was not considered a new exacerbation.
Time Frame: Baseline (Day 1) to Week 24
Population: ITT population included all participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg | Placebo
Number analyzed (Participants) | 82 | 87 | 87
Participants | 26 | 29 | 42

ADVERSE EVENTS:
Time Frame: Baseline to Week 28 (End of study visit)
Description: Safety population included all participants who received at least one dose of study treatment.
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/81 | 1/89 | 0/85
Serious Adverse Events (participants affected / at risk) | 11/81 | 10/89 | 19/85
Other Adverse Events (participants affected / at risk) | 47/81 | 43/89 | 33/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brensocatib 10 mg (N=81) | Brensocatib 25 mg (N=89) | Placebo (N=85)
Infective exacerbation of bronchiectasis (Infections and infestations) | 5 | 4 | 9
Pneumonia (Infections and infestations) | 0 | 4 | 3
Bronchitis (Infections and infestations) | 1 | 0 | 0
Aspergilloma (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brensocatib 10 mg (N=81) | Brensocatib 25 mg (N=89) | Placebo (N=85)
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 9
Periodontal disease (Gastrointestinal disorders) | 2 | 5 | 0
Fatigue (General disorders) | 3 | 7 | 6
Upper respiratory tract infection (Infections and infestations) | 6 | 4 | 4
Sinusitis (Infections and infestations) | 5 | 4 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1 | 1
Headache (Nervous system disorders) | 8 | 12 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 12 | 10
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 1
Hypertension (Vascular disorders) | 2 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT03218917/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT03218917/SAP_001.pdf